CLINICAL TRIAL: NCT01914705
Title: Landmark vs. Ultrasound Guided Subclavian Central Venous Catheter Placement in the Emergency Department
Brief Title: Landmark vs. Ultrasound Guided SCVC in the ED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Too few patients who met enrollment criteria.
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Manager, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11/12/VA01
Record Dates: First submitted 2013-07-31; First posted 2013-08-02 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-07

CONDITIONS: Hypotensive
Keywords: Landmark; Ultrasound; central venous catheter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Landmark Procedure (Active Comparator): Using Landmarks to guide SCVC placement
  Interventions: Procedure: Landmark Procedure
- Ultrasound Guided Procedure (Active Comparator): Using ultrasound to guide SCVC placement
  Interventions: Procedure: Ultrasound Guided Procedure

INTERVENTIONS:
Procedure: Landmark Procedure — Using Landmarks to guide SCVC placement
  Arms: Landmark Procedure
Procedure: Ultrasound Guided Procedure — Using ultrasound to guide SCVC placement
  Arms: Ultrasound Guided Procedure

SUMMARY:
The objective of the study is to investigate whether or not there will be a significant difference between landmark vs. ultrasound guided approach during Subclavian Central Venous Catheter (SCVC) placement in terms of the success rate, the time it takes to perform the procedure and the complication rate. By using ultrasound to identify anatomical structures that are not seen during the landmark approach, the investigators hypothesize that both the procedural time and the complication rate of ultrasound guided approach should be lower than the landmark approach. The investigators hypothesize that the success rate will be higher in the ultrasound group.

DETAILED DESCRIPTION:
Placement of a central venous catheter (CVC) is a common critical care procedure performed by emergency physicians in the Emergency Department (ED.) Numerous studies have shown that physicians are able to reduce the time required, the complication rates, and the number of attempts, and to increase the overall success of CVC placement with the use of ultrasound guidance. Thus, ultrasound guided CVC placement is being increasingly utilized in the ED. The investigators propose a study to investigate the utility of ultrasound guidance for placement of subclavian CVC (SCVC) in the ED.

Currently there are numerous studies, including prospective randomized trials, comparing landmark and ultrasound guided placements of Internal Jugular(IJ) and Femoral CVC, both in the ED and in the ICU settings. However, there has not yet been a prospective randomized trial that has similarly looked at SCVC placement in the ED setting. There are a few studies looking at ultrasound guided SCVC placement performed in critical care settings, but these trials had methodological limitations. Recently, a large (401 patients), randomized, prospective study from an ICU in Greece was published in which the landmark approach was compared to ultrasound guided SCVC placement. The authors found that ultrasound guided SCVC was superior to the landmark approach in success rate, time to cannulation, and complication rates.

The investigators would like to conduct a similar prospective randomized study in the ED, in which the investigators compare the success rate, the procedural times and the complication rates between landmark and real-time ultrasound guided approaches to SCVC placement. In contrast to the recent Greek study, this study will involve a different patient population. The Greek study only looked at ventilated ICU patients, and this study will look at adult patients in the ED setting.

Once an independent clinical decision has been reached to place an SCVC by the ED attending physician, the study investigators will be contacted to enroll the patient. Patients will be randomly assigned to receive either landmark or ultrasound guided SCVC placement. In the ultrasound guidance group, a two person technique will be utilized in which the ultrasound machine will be operated by one of the investigating physicians, and the catheter will be placed by the ED physician caring for the patient. The investigators will employ real time ultrasound guidance using both the transverse and longitudinal views to help direct the needle to the vein. Once the vascular structures are identified on ultrasound by the investigating physician, the physician placing the SCVC will be directed to puncture the skin at the optimal location as determined by the investigating physician. Ultrasound will be used throughout the entire procedure to cannulate the underlying vein. In the landmark group, the SCVC will be placed using anatomic landmarks to locate the puncture site by the physicians working clinically in the ED. The Seldinger technique used for SCVC placement is the same for both the landmark and ultrasound guided approaches.

Using a stopwatch, the investigating physician will document a "Begin Time" just after the patient and the equipment have been prepped under full sterile precautions. In both groups, the timer would start at the same point in time - - when the needle is ready to puncture the skin. Complications will also be noted by the investigating physician during and after the SCVC placement, including number of puncture attempts, success/failure of blood return from the SCVC ports, occurrence of catheter tip misplacement, arterial puncture, and incidence of hematoma, hemothorax, or pneumothorax. As per routine protocol, a post-procedure chest x-ray will be obtained and will be reviewed for evidence of complications. The final Radiology Attending interpretation of the chest xray will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Department Adult Patients
* Need placement of subclavian central venous catheter

Exclusion Criteria:

* Patients with known coagulopathy
* Patients with history of subclavian thrombosis
* Patients with history of vascular injury
* Pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Success Rate | 30 minutes
  Measure whether or not the physician was able to successfully place the subclavian central venous catheter (SCVC).

SECONDARY OUTCOMES:
Procedure Time | 30 minutes
  Measure the time it takes the physician to perform the subclavian catheter placement procedure.

OTHER OUTCOMES:
Complication Rate | 30 minutes
  Measure the complication rate of the physician's procedure of subclavian central venous catheter placement.

CONTACTS AND LOCATIONS:
Overall Officials: John Marshall, MD, Study Chair — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States